CLINICAL TRIAL: NCT01092039
Title: XIGO Effectiveness Study: An Investigation of the Safety and Efficacy of Oral XIGO Tablets on Patients Diagnosed With the Common Cold
Brief Title: Safety and Efficacy Study of Oral XIGO Tablets to Treat The Common Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xigo Health LLC (Industry)
Responsible Party: Rudy Beeck, CEO, XIGO Health, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XIGO-001
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2011-06

CONDITIONS: Common Cold
Keywords: Common Cold; Cold Virus; Feeling sick; Influenza
MeSH Terms: conditions — Common Cold; Nausea; Influenza, Human | interventions — Lactoferrin; Glutamine; beta-Glucans

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XIGO pill (Experimental): Oral Xigo tablet
  Interventions: Dietary Supplement: lactoferrin, L-Glutamine and beta-glucans
- Placebo (Placebo Comparator): Oral placebo tablet
  Interventions: Dietary Supplement: lactoferrin, L-Glutamine and beta-glucans; Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: lactoferrin, L-Glutamine and beta-glucans — Subject will be given XIGO pills or placebo. two tablets to be taken by mouth 3 times per day.
Dietary Supplement: Placebo Comparator — Subject will be given placebo comparator of two tablets to be taken by mouth 3 times per day.
  Arms: Placebo

SUMMARY:
The purpose of the study will be to assess the efficacy and safety of XIGO administered orally, three times a day, compared with placebo in patients with the common cold.

DETAILED DESCRIPTION:
The common cold is one of the most frequent human illnesses and has been shown to result in significant morbidity and economic loss. At the present time no truly effective therapy is available. Therapeutic interventions with compounds such as zinc have been found to be helpful however well reported side-effects have prevented its extensive use.

Based on several years of anecdotal clinical evidence which has shown that XIGO is effective in alleviating the symptoms of the common cold-the findings of which are supported by competent and reliable evidence from in vivo and in vitro and clinical trials studies on each of the individual active ingredients of the formulation, it has been proposed that XIGO, when administered orally, has a direct stimulatory effect on multiple components of the immune system. It is proposed that this stimulation increases both the immune cell population as well as its functionality and this will be observed in cells and molecules from both the innate and adaptive responses.

ELIGIBILITY:
Inclusion Criteria:

* Must be in good health in the clinical judgment of the investigator, other than cold symptoms
* Must have a cumulative score of 2 or higher, but not larger than 6, with symptom severity rated as 0=absent, 1=mild, 2= moderate, or 3=severe for each of the eight symptoms: sneezing, nasal discharge, nasal obstruction, sore throat, cough, headache, malaise and chillness. At least one of the first four "cold specific" symptoms must be present, and none of these symptoms can have been present for more than 12 hours.
* Must enter trial within 12 hours of symptoms onset.
* Aged 18-50 years, (inclusive), at visit 1.
* Subjects must understand and sign and date an informed consent form prior to any study related procedures being performed.
* Subjects must be capable of understanding and following directions.

Exclusion Criteria:

* Subjects taking medications, other than birth control, which, in the opinion of the investigator, could influence the purpose, integrity or outcome of the trial.
* Pre-menopausal women (last menstruation <=1 year prior to ICF) who are nursing or pregnant or are of child-bearing potential and, in the opinion of the investigator, are not practicing an acceptable method of birth control, or do not plan to continue using method throughout the study.
* A history of adverse reactions to OTC drugs or other personal care products.
* Subjects who have used systemic steroids for at least 6 weeks prior to trial initiation or during the trial.
* A medical history of autoimmune disease, including Type 1 or Type 2 diabetes or HIV.
* Treatment with immunosuppressive drugs with the exception of cyclosporine for keratitis sicca.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Severity of cold symptoms over 7 days. | 7 days post dose
  The primary outcome measure will be to assess the severity of the typical interrelated common cold symptoms, over the first seven days of observation period, with the first day being the 24 hour period after first dose of treatment, using the patient/subject completion of the Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21).

SECONDARY OUTCOMES:
Severity of Cold Symptoms over 14 days | Over 14 day observation period
  The secondary outcome measures will be to assess the severity of the typical interrelated common cold symptoms, over the fourteen days of observation period, with the first day being 24 hours after first dose of treatment, using the patient/subject completion of the WURSS-21.
Assess time to resolution | 14 days post dose
  This secondary outcome is to assess the time to resolution of the typical interrelated common cold symptoms, with resolution deemed to occur when participant reports being "not sick" for two days in a row
Percentage of patients with unresolved symptoms | 14 days post dose
  This secondary outcome is to assess the % of patients with clinically unresolved symptoms at day 14, as accessed by the attending investigator. This will include secondary complications such as rhinitis, sinusitis, lower respiratory tract infections and asthma exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory G Allen J.R., D.O., Principal Investigator — NECCR/ IMCA LLC
Locations (1):
- Neccr/Imca Llc, Fall River, Massachusetts, United States